CLINICAL TRIAL: NCT04465903
Title: Validity and Reliability of the Turkish Version of the Sydney Swallow Questionnaire (SSQ-T)
Brief Title: Validity and Reliability of the Turkish Version of the Sydney Swallow Questionnaire
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Yavuz Atar, Associate Professor, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 298
Record Dates: First submitted 2020-07-03; First posted 2020-07-10 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Dysphagia, Oropharyngeal; Swallowing Disorder; Validation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysphagia patients: The first group consists of 85 dysphagia patients who have at least six months of dysphagia complaints. The participants will given the Turkish version of Sydney Swallow questionnaire (SSQ-T), consisted of 17 questions, eating assessment tool-10 and two scales evaluated with FEES. After the two weeks, 30 participants will given the SSQ-T for sampling.
  Interventions: Other: Turkish Version of Sydney Swallow Questionnaire
- Healthy adults: The second group consists of 85 healty participants will given the SSQ-T consists of 17 questions, eating assessment tool-10.
  Interventions: Other: Turkish Version of Sydney Swallow Questionnaire

INTERVENTIONS:
Other: Turkish Version of Sydney Swallow Questionnaire — The Turkish Version of Sydney Swallow Questionnaire consists of 17 questions related with dysphagia.

SUMMARY:
Purpose of the study is the validity and reliability of the Turkish version of the Sydney Swallow Questionnaire (SSQ-T), so that it would be used as an assessment tool for Turkish dysphagia patients. Despite being translated and validated in many languages, there is no validated Turkish version of SSQ to measure the severity of oropharyngeal dysphagia.

DETAILED DESCRIPTION:
The swallow function is a multidirectional process that depends on complex neuro-muscular network. The function can be evaluated using instrumental, such as fibreoptic endoscopic evaluation of swallowing (FEES), videofluoroscopy, or well structured questionnaires. There are many questionnaire and scales for assessment of swallow but very few have been validated. The study will assess the construct validity and reliability of the Turkish version of Self-report Symptom Inventory as known as Sydney Swallow Questionnaire. The investigators developed the Turkish version of this questionnaire (SSQ-T), according to the cross-cultural adaptation guidelines. Two translators translated the SSQ into Turkish and a native English language speaker reverse-translated it into English. The back translation was sent to the original author for proofreading. The SSQ questionnaire consisted of 17 basic questions related with dysphagia symptoms.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Able to speak, read, understand and write in Turkish
* History of dysphagia during 6 months
* Age between 18-80 years

Group 2:

* Able to speak, read, understand and write in Turkish
* Healthy adults
* Age between 18-80 years old.

Exclusion Criteria:

* Mental disorders
* Cognitive limitations
* Able not to speak, read, understand and write in Turkish
* Underwent any surgery last a month
* Underwent laryngectomy/neck dissection/tracheostomy/neck radiotherapy
* Pregnancy
* Malignancies
* Out of age 18-80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with oropharyngeal dysphagia and healthy adults
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Turkish Version of Sydney Swallow Questionnaire | Baseline
  Turkish version of the questionnaire consists of 17 questions about dysphagia and swallowing functions and dysphagia consequences during patients at least six months and healty subjects. The minimum score is 0 and maximum score is 1700. The lower scores mean a normal swallowing function, higher scores mean worst oropharyngeal swallowing functions.
Turkish Version of Sydney Swallow Questionnaire | 2 weeks
  Turkish version of the questionnaire consists of 17 questions about dysphagia and swallowing functions and dysphagia consequences during patients at least six months. The minimum score is 0 and maximum score is 1700. The lower scores mean is a normal swallowing function, higher scores mean is worst oropharyngeal swallowing functions.

SECONDARY OUTCOMES:
Eating Assessment Tool | Baseline
  The Turkish validated questionnaire consists of 10 questions that scores are from 0 to 40. Low score is better, higher score is worse.
Penetration and aspiration scale | Baseline
  The scale consists of 8 levels for assessment of penetration and aspiration. The scores are from 0 to 8. Low score is better, higher score is worse.
YALE scale of pharyngeal residue | Baseline
  The scale consists of 5 assessment units for pharyngeal residue. The scores are from 1 to 5. Low score is better, higher score is worse.

OTHER OUTCOMES:
Subject demographics | Baseline
  The median values of age and ratio of gender in all groups

CONTACTS AND LOCATIONS:
Overall Officials: Melis Ece Arkan Ararat, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization; Ugur Uygan, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arenaz Bua B, Bulow M. Validation in Swedish of Sydney swallow questionnaire. BMC Res Notes. 2014 Oct 21;7:742. doi: 10.1186/1756-0500-7-742. PMID 25330714
- [Result] Audag N, Goubau C, Danse E, Vandervelde L, Liistro G, Toussaint M, Reychler G. Validation and Reliability of the French Version of the Sydney Swallow Questionnaire. Dysphagia. 2019 Aug;34(4):556-566. doi: 10.1007/s00455-019-09978-9. Epub 2019 Feb 1. PMID 30707281
- [Result] Dwivedi RC, St Rose S, Chisholm EJ, Georgalas C, Bisase B, Amen F, Kerawala CJ, Clarke PM, Nutting CM, Rhys-Evans PH, Harrington KJ, Kazi R. Evaluation of swallowing by Sydney Swallow Questionnaire (SSQ) in oral and oropharyngeal cancer patients treated with primary surgery. Dysphagia. 2012 Dec;27(4):491-7. doi: 10.1007/s00455-012-9395-z. Epub 2012 Feb 21. PMID 22350113
- [Result] Wallace KL, Middleton S, Cook IJ. Development and validation of a self-report symptom inventory to assess the severity of oral-pharyngeal dysphagia. Gastroenterology. 2000 Apr;118(4):678-87. doi: 10.1016/s0016-5085(00)70137-5. PMID 10734019